CLINICAL TRIAL: NCT05303402
Title: A Phase IIb/III, Open Label, Single Arm, Multi-centre, Trial to Assess the Immunogenicity and Safety of an Additional Dose Vaccination With a Recombinant Protein RBD Fusion Heterodimer Candidate (PHH-1V) Against SARS-CoV-2, in Adults With Pre-existing Immunosuppressive Conditions Vaccinated Against COVID-19
Brief Title: A Phase IIb/III Clinical Trial to Assess Safety and Immunogenicity of a COVID-19 Vaccine Booster Dose in Immunosupressed Adults.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hipra Scientific, S.L.U (Industry)
Collaborators: Veristat, Inc. (Other); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Asphalion (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HIPRA-HH-4
Record Dates: First submitted 2022-03-28; First posted 2022-03-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19 | interventions — HIPRA COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: COVID-19 Vaccine HIPRA 40 mcg/dose (Experimental): Intramuscular injection of HIPRA's COVID-19 vaccine, consisting of 40 mcg/dose.
  Interventions: Biological: PHH-1V

INTERVENTIONS:
Biological: PHH-1V — COVID-19 Vaccine HIPRA, 40 mcg/dose

SUMMARY:
A phase IIb/III, open label, single arm, multi-centre, trial to assess the immunogenicity and safety of an additional dose vaccination with a recombinant protein RBD fusion heterodimer candidate (PHH-1V) against SARS-CoV-2, in adults with pre-existing immunosuppressive conditions vaccinated against COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Male, female or transgender, ≥ 18 years old at Day 0.
* Provide inform consent form
* Participant who has:
* 3 doses of mRNA vaccines
* 2 doses of mRNA vaccines and previous COVID-19 infection
* 2 doses of Coronavac and 1 Comirnaty, or, 1 Coronavac and 2 Comirnaty
* Participant who has:
* HIV infection with CD4 Tcells counts <400
* Primary antibody deficiency disorders
* Kidney disease on dialysis
* Kidney transplant at least >1 year
* Auto Immune Disease (AID) in treatment with rituximab
* For a female of childbearing potential, to have a negative pregnancy test at Day 0
* Use of any of these contraception:
* Female: hormonal contraception, intrauterine device, vasectomized partner, sexual abstinence, condom.
* Male: Vasectomized participant, sexual abstinence, condom.

Exclusion Criteria:

* History of anaphylaxis to any prior vaccine
* Participants has received or plans to receive live attenuated vaccines, other not live vaccines, or Vaxzevria or Janssen vaccines.
* Pregnant or breast-feeding at Day 0.
* A confirmed COVID-19 diagnose <90 days prior to vaccination day 0.
* A clinically significant acute illness or fever at screening or 48h before day 0.
* Participant had a surgery requiring hospitalisation and has not received the hospital discharge.
* Participant has an ongoing severe and non-stable psychiatric condition
* Participant has a problematic or risky use of substances including alcohol
* Participant has a bleeding disorder that contraindicates intramuscular injection
* Participant suffering from post-acute COVID-19 syndrome / long COVID
* Participant received any immunotherapy to prevent/treat COVID-19 in the last 90 days
* Participant is already participating in another research involving drug, biologics or device
* Participant has donated ≥450 ml of blood products within 12 weeks before screening
* Participant has any medical condition and/or finding that in the investigator opinion might increase participant risk, interfere with the study or impair interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity against Omicron, Beta, Delta at Day 0 and Day 14 | Day 0 and Day 14
  Changes in neutralising antibodies measured by pseudovirus (or live virus for the HIV cohort*) neutralization against Omicron, Beta and Delta any other relevant Variants of Concern (VOC) in the epidemiologic moment, at Baseline and at Day 14 after administration of HIPRA's vaccine (PHH-1V).

SECONDARY OUTCOMES:
Immunogenicity against Omicron, Beta, Delta at Day 91, Day 182 and Day 365 | Day 91, Day 182 and Day 365
  1. To determine and compare the changes of the immunogenicity measured by pseudovirus (or live virus for the HIV cohort) neutralization against Omicron, Beta and Delta and any other relevant Variants of Concern (VOC) in the epidemiologic moment at Days, 91, 182 and 365, after administration of HIPRA's vaccine (PHH-1V).
Total antibodies | Day 0, Day 14, Day 91, Day 182, Day 365
  To evaluate the immunogenicity measured by means of total antibody against Receptor Binding Domain of the Spike protein of SARS-CoV-2 quantification, measured by an electrochemiluminescence immunoassay (ECLIA) at Baseline and at Days 14, 91, 182 and 365 after administration of HIPRA's vaccine (PHH-1V).
Safety and tolerability of the booster vaccine | Day 0, Day 14, Day 91, Day 182, Day 365
  To assess the safety and tolerability of PHH-1V as an additional dose in adult individuals with pre-existing immunosuppressive conditions

OTHER OUTCOMES:
Number of SARS-CoV-2 infections | Day 0, Day 14, Day 91, Day 182, Day 365
  Number of participants with SARS-CoV-2 infections ≥14 days after PHH-1V administration.
Number of SARS-CoV-2 severe infections (Severe cases are considered as any episode of COVID-19 requiring ≥ 24hrs of hospitalization.) | Day 0, Day 14, Day 91, Day 182, Day 365
  Number of COVID-19 severe infections ≥14 days after PHH-1V administration.
Celular immunity | Day 0, Day 14, Day 91, Day 182, Day 365
  Antibody IgG subclasses titre usage and avidity of humoral immunity at Baseline and Days 14, 91, 182 and 365.
T-cell cellullar immunity | Day 0, Day 14, Day 91, Day 182, Day 365
  T-cell mediated phenotype polyclonality with potential cross-reactivity capacity and gene-expression profiles against the SARS-CoV-2 Spike & RBD proteins at Baseline and at Days 14, 91, 182 and 365 in a subset of 50% of participants.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (3):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Josep Trueta, Girona, Girona
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty Hospitals, Ankara, Ankara
  - Ankara University Medical Faculty Hospitals, Ankara, Ankara
  - Koc University Hospital, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: No